CLINICAL TRIAL: NCT04200781
Title: A Randomized, Controlled, Double-blind, Multi-center Clinical Study of Shengdi Dahuang Decoction in the Treatment of Acute Hemorrhagic Stroke
Brief Title: Clinical Evaluation of Shengdi Dahuang Decoction in the Treatment of Acute Hemorrhagic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Xiaofei Yu, Clinical Professor, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19401972800
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Hemorrhagic Stroke
Keywords: acute hemorrhagic stroke; Shengdi Dahuang Decoction
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shengdi Dahuang Decoction (Experimental): To clarify the clinical effects of Shengdi Dahuang Decoction in the treatment of acute hemorrhagic stroke and to explore the possible mechanism. Participants will take the granules of Shengdi Dahuang Decoction that contains 15 grams of rehmannia and 5 grams of rhubarb, one pack per time, twice a day for 7 days.
  Interventions: Drug: Granules of Shengdi Dahuang Decoction
- Placebo (Placebo Comparator): To explore the effective clinical therapy in acute hemorrhagic stroke. Participants will take placebo contains 2% rehmannia and rhubarb, one pack per time, twice a day for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granules of Shengdi Dahuang Decoction — Shengdi Dahuang Decoction contains Shengdi (rehmannia) and Dahuang ( rhubarb). Each pack of the granules of Shengdi Dahuang Decoction contains 15 grams of rehmannia and 5 grams of rhubarb.
  Other Names: Chinese Herbal Compound
  Arms: Shengdi Dahuang Decoction
Drug: Placebo — Placebo granules has the same appearence, weight, shape and color as the experimental drug.
  Other Names: Placebo of Chinese Herbal Compound
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Shengdi Dahuang Decoction in the treatment of acute hemorrhagic stroke by the randomized, controlled, double-blind, multi-center trial design project.

DETAILED DESCRIPTION:
The main purpose of the study is to observe the clinical efficacy and safety of Shengdi Dahuang Decoction in the treatment of acute hemorrhagic stroke. This project is funded by Science and Technology Commission of Shanghai Municipality and will be carried out in 5 hospitals. Investigators will recruit 464 participants who meet the inclusion criteria and agree to participate in the research. Participants will be randomly assigned into experimental or placebo group. Granules of Shengdi Decoction is the therapeutic drug used in the experimental group. Each pack of the test drug contains 15 grams of rehmannia and 5 grams of rhubarb. While for the placebo group, each pack contains 2% rehmannia and rhubarb. Participants will receive a follow-up observation in the following 90 days. Modified Rankin Scale score (mRS), the mortality rate on day 7 and day 90 after treatment, National Institute of Health Stroke Scale (NIHSS), expansion rate of hematoma, the degree of edema and the expressions of inflammatory indicators will be detected to evaluate the clinical efficacy of Shengdi Dahuang Decoction.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of acute intracerebral hemorrhage；
2. CT scan reveals cerebral parenchymal hemorrhage and the volume of hematoma is <80ml;
3. The time from onset to confirmed diagnosis by CT scan is within 4 hours;
4. Enrolled and receive treatment within 12 hours from onset;
5. Age ≥18 years old;
6. Obtain approval from the patient or family members.

Exclusion Criteria:

1. The time from onset to confirmed diagnosis by CT scan is over 4 hours;
2. CT scan indicate that the sites of hemorrhage are in the cerebellum, brainstem and ventricle (note: in case of cerebral parenchymal hemorrhage combined with ventricular hemorrhage, patients will be excluded if the volume of ventricular hemorrhage is the larger one);
3. The volume of hematoma is above 80ml;
4. Glasgow Coma Scale (GCS) is ≤ 5 points;
5. The time from onset to confirmed diagnosis is over 12 hours;
6. Have a surgical treatment planning within 24 hours;
7. Cerebral hemorrhage caused by trauma, arteriovenous malformation, thrombolytic therapy, anticoagulant therapy or other reasons;
8. Patients with disabilities before onset (modified mRS score > 2);
9. Patients with severe primary diseases of the heart, lung, liver, kidney, endocrine systems or hematopoietic system;
10. Patients who have participated in other clinical trials within the past 1 month;
11. Pregnant or nursing women;
12. Allergic constitution (allergic to more than two kinds of food or medications).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Disability rate | 90 days
  Modified Rankin Scale score (mRS) will be graded on the 90th day after onset (mRS score ranges from 0 point (no symptoms at all) to 5 points (severe disability)).
Mortality rate on the 7th day | 7 days
  The proportion of deaths (mortality rate, %) in different groups on 7th day after treatment will be compared.

SECONDARY OUTCOMES:
Mortality rate on the 90th day | 90 days
  The proportion of deaths (mortality rate, %) in different groups on 90th day after treatment will be compared.
Severity of neurological deficit | 7 days
  National Institute of Health Stroke Scale (NIHSS) will be used to assess the severity of neurological deficit on the 7th day after treatment. NIHSS score ranges from 0 point to 42 points. More severe neurological deficit could be observed in participants with the higher score.
The proportion of hematoma enlargement cases | 24 hours
  All participants will reexamine the skull CT scan 24 hours after onset. The volume of hematoma (ml) increases more than 6ml or 33% relative increment than original volume is defined as the expansion of hematoma. The proportion of hematoma enlargement cases (%) will be compared between different groups.
Severity of edema | 7 days
  All participants will reexamine the skull CT scan on the 7th day after treatment. The volume (ml) of edema and hematoma will be calculated respectively. The ratio of edema volume and hematoma volume represents the severity of edema.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Yu, Study Chair — Shuguang Hospital affiliated with Shanghai University of TCM
Locations (5):
- China (5):
  - Shanghai seventh People's Hospital, Seventh People's Hospital of Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shuguang Hospital affiliated with Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arima H, Heeley E, Delcourt C, Hirakawa Y, Wang X, Woodward M, Robinson T, Stapf C, Parsons M, Lavados PM, Huang Y, Wang J, Chalmers J, Anderson CS; INTERACT2 Investigators; INTERACT2 Investigators. Optimal achieved blood pressure in acute intracerebral hemorrhage: INTERACT2. Neurology. 2015 Feb 3;84(5):464-71. doi: 10.1212/WNL.0000000000001205. Epub 2014 Dec 31. PMID 25552575
- [Result] Cai M, Yu Z, Zhang W, Yang L, Xiang J, Zhang J, Zhang Z, Wu T, Li X, Fu M, Bao X, Yu X, Cai D. Sheng-Di-Da-Huang Decoction Inhibited Inflammation Expressed in Microglia after Intracerebral Hemorrhage in Rats. Evid Based Complement Alternat Med. 2018 Oct 18;2018:6470534. doi: 10.1155/2018/6470534. eCollection 2018. PMID 30498516
- [Result] Chang JJ, Emanuel BA, Mack WJ, Tsivgoulis G, Alexandrov AV. Matrix metalloproteinase-9: dual role and temporal profile in intracerebral hemorrhage. J Stroke Cerebrovasc Dis. 2014 Nov-Dec;23(10):2498-2505. doi: 10.1016/j.jstrokecerebrovasdis.2014.07.005. Epub 2014 Oct 11. PMID 25306400
- [Result] Behrouz R, Azarpazhooh MR, Godoy DA, Hoffmann MW, Masotti L, Parry-Jones AR, Popa-Wagner A, Schreuder FH, Slevin MA, Smith CJ, Di Napoli M; MNEMONICH Steering Committee. The Multi-National survey on Epidemiology, Morbidity, and Outcomes iN Intracerebral Haemorrhage (MNEMONICH). Int J Stroke. 2015 Dec;10(8):E86. doi: 10.1111/ijs.12629. No abstract available. PMID 26745705
- [Result] Cordonnier C, Demchuk A, Ziai W, Anderson CS. Intracerebral haemorrhage: current approaches to acute management. Lancet. 2018 Oct 6;392(10154):1257-1268. doi: 10.1016/S0140-6736(18)31878-6. PMID 30319113
- [Result] Ding R, Chen Y, Yang S, Deng X, Fu Z, Feng L, Cai Y, Du M, Zhou Y, Tang Y. Blood-brain barrier disruption induced by hemoglobin in vivo: Involvement of up-regulation of nitric oxide synthase and peroxynitrite formation. Brain Res. 2014 Jul 7;1571:25-38. doi: 10.1016/j.brainres.2014.04.042. Epub 2014 May 9. PMID 24814387
- [Result] Flower O, Smith M. The acute management of intracerebral hemorrhage. Curr Opin Crit Care. 2011 Apr;17(2):106-14. doi: 10.1097/MCC.0b013e328342f823. PMID 21169826
- [Result] Garg R, Biller J. Recent advances in spontaneous intracerebral hemorrhage. F1000Res. 2019 Mar 18;8:F1000 Faculty Rev-302. doi: 10.12688/f1000research.16357.1. eCollection 2019. PMID 30906532
- [Result] Geng X, Ren C, Wang T, Fu P, Luo Y, Liu X, Yan F, Ling F, Jia J, Du H, Ji X, Ding Y. Effect of remote ischemic postconditioning on an intracerebral hemorrhage stroke model in rats. Neurol Res. 2012 Mar;34(2):143-8. doi: 10.1179/1743132811Y.0000000073. Epub 2012 Jan 13. PMID 22333136
- [Result] Gregson BA, Mitchell P, Mendelow AD. Surgical Decision Making in Brain Hemorrhage. Stroke. 2019 May;50(5):1108-1115. doi: 10.1161/STROKEAHA.118.022694. PMID 30932784
- [Result] Hanley DF, Lane K, McBee N, Ziai W, Tuhrim S, Lees KR, Dawson J, Gandhi D, Ullman N, Mould WA, Mayo SW, Mendelow AD, Gregson B, Butcher K, Vespa P, Wright DW, Kase CS, Carhuapoma JR, Keyl PM, Diener-West M, Muschelli J, Betz JF, Thompson CB, Sugar EA, Yenokyan G, Janis S, John S, Harnof S, Lopez GA, Aldrich EF, Harrigan MR, Ansari S, Jallo J, Caron JL, LeDoux D, Adeoye O, Zuccarello M, Adams HP Jr, Rosenblum M, Thompson RE, Awad IA; CLEAR III Investigators. Thrombolytic removal of intraventricular haemorrhage in treatment of severe stroke: results of the randomised, multicentre, multiregion, placebo-controlled CLEAR III trial. Lancet. 2017 Feb 11;389(10069):603-611. doi: 10.1016/S0140-6736(16)32410-2. Epub 2017 Jan 10. PMID 28081952
- [Result] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Result] Hao S, Wang B. Editorial: Review on Intracerebral Haemorrhage: Multidisciplinary Approaches to the Injury Mechanism Analysis and Therapeutic Strategies. Curr Pharm Des. 2017;23(15):2159-2160. doi: 10.2174/1381612823999170307150448. No abstract available. PMID 28703081
- [Result] Mayer SA, Brun NC, Begtrup K, Broderick J, Davis S, Diringer MN, Skolnick BE, Steiner T; FAST Trial Investigators. Efficacy and safety of recombinant activated factor VII for acute intracerebral hemorrhage. N Engl J Med. 2008 May 15;358(20):2127-37. doi: 10.1056/NEJMoa0707534. PMID 18480205
- [Result] Morotti A, Brouwers HB, Romero JM, Jessel MJ, Vashkevich A, Schwab K, Afzal MR, Cassarly C, Greenberg SM, Martin RH, Qureshi AI, Rosand J, Goldstein JN; Antihypertensive Treatment of Acute Cerebral Hemorrhage II and Neurological Emergencies Treatment Trials Investigators. Intensive Blood Pressure Reduction and Spot Sign in Intracerebral Hemorrhage: A Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2017 Aug 1;74(8):950-960. doi: 10.1001/jamaneurol.2017.1014. PMID 28628707
- [Result] Rivest S. Regulation of innate immune responses in the brain. Nat Rev Immunol. 2009 Jun;9(6):429-39. doi: 10.1038/nri2565. PMID 19461673
- [Result] Selim M, Sheth KN. Perihematoma edema: a potential translational target in intracerebral hemorrhage? Transl Stroke Res. 2015 Apr;6(2):104-6. doi: 10.1007/s12975-015-0389-7. Epub 2015 Feb 20. No abstract available. PMID 25693976
- [Result] Sprigg N, Flaherty K, Appleton JP, Al-Shahi Salman R, Bereczki D, Beridze M, Christensen H, Ciccone A, Collins R, Czlonkowska A, Dineen RA, Duley L, Egea-Guerrero JJ, England TJ, Krishnan K, Laska AC, Law ZK, Ozturk S, Pocock SJ, Roberts I, Robinson TG, Roffe C, Seiffge D, Scutt P, Thanabalan J, Werring D, Whynes D, Bath PM; TICH-2 Investigators. Tranexamic acid for hyperacute primary IntraCerebral Haemorrhage (TICH-2): an international randomised, placebo-controlled, phase 3 superiority trial. Lancet. 2018 May 26;391(10135):2107-2115. doi: 10.1016/S0140-6736(18)31033-X. Epub 2018 May 16. PMID 29778325
- [Result] Toyoda K, Grotta JC. Seeking best medical treatment for hyperacute intracerebral hemorrhage. Neurology. 2015 Feb 3;84(5):444-5. doi: 10.1212/WNL.0000000000001221. Epub 2014 Dec 31. No abstract available. PMID 25552577
- [Result] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Result] Wang J. Preclinical and clinical research on inflammation after intracerebral hemorrhage. Prog Neurobiol. 2010 Dec;92(4):463-77. doi: 10.1016/j.pneurobio.2010.08.001. Epub 2010 Aug 14. PMID 20713126
- [Derived] Sun Z, Zhou X, Xiang J, Wang F, Han Y, Guo Y, Zhang Z, Gong F, Wang M, Liu D, Pan W, Tang H, Li T, Zhang J, Jiang S, Huang J, Yu X. Treatment of acute intracerebral haemorrhage with a Chinese herbal formula (Shengdi Dahuang Decoction): a multicentre, double-blind, randomised, placebo-controlled trial. Stroke Vasc Neurol. 2025 Aug 2:svn-2024-003931. doi: 10.1136/svn-2024-003931. Online ahead of print. PMID 40752894